CLINICAL TRIAL: NCT06994338
Title: Phase II Evaluation of Tirzepatide in Adults With Alcohol Use Disorder and Overweight or Obesity
Brief Title: Tirzepatide for Alcohol Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christian Hendershot, Professor and Director of Clinical Research, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-25-00273; 1R21AA031892-01 (NIH)
Record Dates: First submitted 2025-05-16; First posted 2025-05-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder; Obesity and Overweight; Alcohol
Keywords: Tirzepatide; GLP-1; Addiction; Alcohol
MeSH Terms: conditions — Alcoholism; Obesity; Overweight; Behavior, Addictive | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental)
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo injections

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide injections (2.5mg, 5.0mg)
  Arms: Tirzepatide
Drug: Placebo injections — Placebo injections
  Arms: Placebo

SUMMARY:
The objective of this Phase 2 randomized controlled trial is to evaluate the effects of weekly tirzepatide (vs. placebo) on alcohol consumption and cardiometabolic outcomes in adults with alcohol use disorder and overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting past-year DSM-5 criteria for AUD with at least moderate severity (≥ 4 symptoms)
2. Average daily consumption of ≥40g (women) / ≥ 60 g (men) per day in the 28 days prior to baseline
3. Body mass index ≥ 27kg/m2
4. Willingness to attend weekly medication visits and complete all study procedures
5. Ability to read and communicate in English
6. Age 21-65
7. Treatment-seeking (i.e., currently seeking assistance to reduce or stop drinking)
8. Stable housing status

Exclusion Criteria:

1. Meeting past-year DSM-5 criteria for another substance use disorder (except tobacco use disorder or mild cannabis use disorder)
2. Recent (past 30 day) self-report of illicit drug use (excluding cannabis) or non-prescribed opioids; or positive urine screen for illicit drugs. A positive screen for opioids will be allowed if the participant is prescribed an opioid replacement therapy medication and can provide documentation.
3. History of significant alcohol withdrawal, as indicated by history of seizure, delirium tremens; history of hospitalization for withdrawal-related symptoms; a CIWA score >9 at assessment; or a baseline score 4+ on the Prediction of Alcohol Withdrawal Severity (PAWS) scale.
4. Recent (past 3 months) engagement in behavioral or pharmacological alcohol use treatment or currently mandated to receive treatment
5. History of chronic or acute pancreatitis
6. History of Type 1 or Type 2 diabetes, or diabetes-related conditions (e.g., diabetic retinopathy), or baseline HbA1C ≥ 6.5%
7. History of suicide attempt or report of current (past 2 weeks) active suicidal ideation
8. Lifetime diagnosis of severe mental illness (e.g., psychosis or bipolar disorder)
9. Evidence of a significant anxiety or depressive disorder that is currently interfering with daily functioning, based on GAD-7 and PHQ-9 scores and physician judgement. (Anxiety or depression are not exclusionary if symptoms are stable/non-interfering with daily activities, or if the participant is receiving treatment, i.e., psychiatric medications have not changed for at least 3 months prior to baseline)
10. Treatment for eating disorder in the past 12 months
11. Report of significant medical, neurological, or psychiatric illness that would preclude safe or full study participation based on the judgement of the study physicians
12. History of known liver disease
13. Elevated serum lipase, amylase, bilirubin, or ALP, ALT, or AST (>3x upper limit of normal range)
14. History of malignant neoplasms in the last 5 years, except for non-melanoma skin cancer
15. Inability to attend weekly clinic visits as scheduled (i.e., based on travel or work schedule)
16. Weight loss > 5% in the 30 days prior to screening
17. Currently enrolled in another clinical trial involving an investigational product
18. Current contact or co-habitation with a current or former participant in the present trial
19. Current co-habitation with a person taking GLP-1RA therapy
20. Planned surgical procedures requiring anesthesia within 90 days post-entry into the study
21. History of treatment with tirzepatide or a GLP-1RA within 6 months of screening
22. Treatment with any weight loss medications (e.g., orlistat, bupropion-naltrexone) or medications known to reduce alcohol consumption (e.g., naltrexone, topiramate, acamprosate, varenicline) in the past 3 months
23. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia (MEN) type I or type II
24. Estimated glomerular filtration rate (eGFR) <60 (indicated impaired kidney function)
25. Use of prescribed or non-prescribed medications that would preclude safe use of tirzepatide in the judgement of the study physicians
26. Known bone, muscle, or wasting conditions (e.g., osteoporosis, sarcopenia) aa. Presence of significant or uncontrolled GI conditions (e.g., GERD) that would interfere with treatment in the judgement of study physicians bb. Any other significant disease, disorder, or finding that in the opinion of the investigator(s) may increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

cc. Currently pregnant or nursing, or inability to adhere to a reliable method of birth control (applies to female participants of childbearing age) dd. Uncontrolled hypertension at baseline, as indicated by an average blood pressure reading of >180/110 after three successive readings ee. History of heart attack or stroke in the 6 months prior to screening ff. A pre-treatment reduction in alcohol consumption to < 40g/day (males) or <20g/day (females) in the interval between baseline screening and randomization

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of heavy drinking days | Last 4 weeks of treatment (Weeks 5-8)
  Number of heavy drinking days (NHDD) during the last four weeks of treatment (treatment Weeks 5-8), as measured by the Timeline Followback interview. NHDD is defined as the total number of days on which participants consumed 5 or more drinks (for men) or 4 or more drinks (for women). The analysis of NHDD will control for baseline NHDD (defined as NHDD in the four weeks preceding treatment).

SECONDARY OUTCOMES:
Drinks per drinking day | Last 4 weeks of treatment (Weeks 5-8)
  Drinks per drinking day (DDD) during the last four weeks of treatment (treatment Weeks 5-8) will be measured by the Timeline Followback interview. DDD is defined as average number of drinks consumed on drinking days. The analysis will control for baseline DDD (defined as DDD in the four weeks preceding treatment).
WHO drinking risk level | Last 4 weeks of treatment (Weeks 5-8)
  WHO risk level is determined based on average grams of daily alcohol consumption, as measured by the Timeline Followback interview. WHO drinking risk level will be measured on a scale from 0-4 (corresponding to abstinence, low, moderate, high, or very high risk). The proportion of participants with a 1-level and 2-level reduction in WHO risk level between baseline (defined as the 28 days prior to the baseline visit) and the final month of treatment (Weeks 5-8) will be computed.
Abstinent days | Last 4 weeks of treatment (Weeks 5-8)
  Abstinent days (proportion of days on which no alcohol consumption is reported) during the last four weeks of treatment (treatment Weeks 5-8) will be measured by the Timeline Followback interview. The analysis will control for baseline (defined as proportion of abstinent days in the four weeks preceding treatment).
Absence of heavy drinking | Last 4 weeks of treatment (Weeks 5-8)
  Absence/remission of heavy drinking in the last month of treatment (treatment Weeks 5-8) will be measured by the Timeline Followback interview. Heavy drinking days are defined as consuming 5 or more drinks (for men) or 4 or more drinks (for women). The change in the proportion of participants with zero heavy drinking days from baseline (defined as the four weeks preceding treatment) to the Weeks 5-8 will be compared across treatment groups.
Alcohol craving | Last 4 weeks of treatment (Weeks 5-8)
  Alcohol craving is measured with the Penn Alcohol Craving Scale (PACS, range: 0-30). Intervention group differences in average weekly craving for the last month of treatment (Weeks 5-8) will be compared. This analysis will control for participants' baseline craving (defined as PACS score assessed at Week 1 prior to the first medication dose).

CONTACTS AND LOCATIONS:
Locations (1):
- Keck School of Medicine, University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes